CLINICAL TRIAL: NCT06529809
Title: Accelerated Brachytherapy Forward Chemo Radiation Therapy (ABC-RT) for Locally-advanced Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202407064; R37CA287204 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Cervical Carcinoma
Keywords: Cervical cancer; Hypofractionated RT; Brachytherapy; Pembrolizumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated Brachytherapy Forward Chemo Radiation Therapy (Experimental): Accelerated Brachytherapy Forward Chemo Radiation Therapy (ABC-RT) combines hypofractionated external beam radiation therapy (EBRT) with concurrent chemotherapy and early upfront, image-guided brachytherapy. In this study, patients start with 2 fractions of brachytherapy prior to initiation of EBRT-based chemoradiotherapy. Total time from treatment planning is approximately 36-42 days.
  Interventions: Radiation: Hypofractionated external beam radiation; Drug: Chemotherapy; Radiation: Image-guided brachytherapy

INTERVENTIONS:
Radiation: Hypofractionated external beam radiation — Central pelvis (19.05 Gy in 15 fractions), nodal basins (40 Gy in 15 fractions), with a simultaneous integrated boost to grossly positive lymph nodes (48 Gy in 15 fractions)
Drug: Chemotherapy — Concurrent chemotherapy are not dictated by the protocol and will follow standard of care guidelines
Radiation: Image-guided brachytherapy — HDR boost 7.3 Gy x 6 fractions

SUMMARY:
The standard treatment for locally advanced cervical cancer is well established as a combination of chemotherapy and radiation, typically over 25-28 daily fractions with the addition of a brachytherapy boost to the primary tumor. An important component to treatment efficacy is overall treatment time. Prolongation of overall treatment time has been shown to lead to worse local control and overall survival; thus, strategies to effectively deliver radiation efficiently is required.

This is a pragmatic feasibility study to determine the impact of upfront brachytherapy combined with hypofractionated external beam radiation for patients with locally advanced cervical cancer (FIGO 2018 stage IB3-IVA) on late gastrointestinal and genitourinary toxicity, oncologic outcomes including recurrence free survival, and systemic and local immune response.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed biopsy proven FIGO (2018) clinical stage IB3-IVA cervical carcinoma.
* Histological diagnosis of squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the cervix
* Candidate for definitive radiation therapy as determined by treating radiation oncologist.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representative may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Any prior pelvic radiotherapy.
* Any prior gynecologic or other pelvic malignancy.
* Any prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for the trial.
* Evidence of metastatic disease outside of the pelvis or para-aortic nodes.
* Previous hysterectomy or planned hysterectomy as part of initial cervical cancer therapy; this includes patients with a prior history of supracervical hysterectomy.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test day of or within 7 days prior to simulation.
* Major surgery ≤ 3 weeks prior to initiating protocol therapy; if a patient has had major surgery prior to 3 weeks, they must have recovered from any surgical effects.
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, or superior vena cava syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Late treatment related grade 3 or greater gastrointestinal and genitourinary adverse events experienced by participant | Between day 91 and 2 year follow-up (estimated to be 2 years and 6 weeks)
  -Must be at least possibly related to RT.

SECONDARY OUTCOMES:
Local recurrence-free survival (LRFS) | Up to 2 year follow-up (estimated to be 2 years and 6 weeks)
  A local recurrence is defined as histologic or radiographic evidence of cancer in the cervix. Local recurrence-free survival is defined as the duration of time from the start of treatment to the time of local recurrence or death, whichever occurs first. The living patients with CR, PR, or SD in the cervix are censored at the corresponding date.
Regional recurrence-free survival (LRFS) | Up to 2 year follow-up (estimated to be 2 years and 6 weeks)
  A regional recurrence is defined as histologic or radiographic evidence of cancer in the pelvic or para-aortic nodes. Regional recurrence-free survival is defined as the duration of time from the start of treatment to the time of regional recurrence or death, whichever occurs first. The living patients with CR, PR, or SD in the pelvis or para-aortic lymph nodes are censored at the corresponding date.
Progression-free survival (PFS) | Up to 2 year follow-up (estimated to be 2 years and 6 weeks)
  Progression- free survival is defined as the duration of time from the start of treatment to progression or death, whichever occurs first. The living patients without progression are censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jessika A Contreras, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of publication.
Access Criteria: Data will be available for investigators whose proposed use of the data has been approved by an independent review committee.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu